CLINICAL TRIAL: NCT06753227
Title: Systematic Assessment of Invasive Versus Echocardiography-derived Transprosthetic Gradients After Transcatheter Aortic Valve Implantation Using Balloon-expandable Transcatheter Heart Valves: the IVEGA-TAVI Study.
Brief Title: Invasive Versus Echocardiography-derived Transvalvular Gradients After TAVI Usign Balloon-expandable Transcatheter Heart Valves.
Acronym: IVEGA-TAVI
Status: Enrolling by invitation | Type: Observational
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-456-S-SB
Record Dates: First submitted 2024-12-22; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: AORTIC VALVE DISEASES; Aortic Stenosis
Keywords: invasive gradients; haemodynamics; aortic valve stenosis; echocardiographic gradients
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with severe aortic valve stenosis requiring transcatheter aortic valve implantation

SUMMARY:
The aim of this prospective registry is to compare invasive versus echocardiography-derived transvalvular gradients before and after TAVI with balloon-expandable THVs.All patients will undergo a transthoracic echocardiogram in the operating room prior to aortic valve implantation. In addition, two catheters (one in the ventricle and one in the aorta) will be used to invasively measure the transvalvular gradient both before and after aortic valve implantation. The invasive measurements will be performed in different positions of the ventricle and aorta simultaneously. At the end of the procedure, aortic gradient measurement by echocardiography shall be performed again. A maximal three months follow-up is expected.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and able to give consent
* Severe symptomatic native aortic valve stenosis with indication for TAVI according to 2021 ESC/EACTS Valvular Heart Disease Guidelines.
* Use of balloon-expandable THV
* Written informed consent

Exclusion Criteria:

* Emergency or urgent treatment indication
* Patients under hemodynamically unstable conditions.
* Previous bioprosthetic aortic valve implantation
* Patient cannot adhere to or complete the trial protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with severe aortic valve stenosis undergoing TAVI with balloon-expandable transcatheter heart valves (THV).
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
To compare transvalvular echocardiographic aortic mean vs. invasive aortic mean gradient after TAVI. | From enrollment to 3 months

SECONDARY OUTCOMES:
To compare transvalvular echocardiographic aortic mean vs. invasive aortic mean gradient before TAVI. | From enrollment to 3 months
To compare pulse-wave Doppler above the aortic valve before and after TAVI | From enrollment to 3 months
To compare pre-ejection period time pre and post TAVI. | From enrollment to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Joner, Professor Dr. med., Study Director — Deutsches Herzzentrum München
Locations (1):
- Deutsches Herzzentrum München, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reddy YNV, Miranda WR, Nishimura RA. Measuring Pressure Gradients After Transcatheter Aortic Valve Implantation: Rethinking the Bernoulli Principle. J Am Heart Assoc. 2021 Oct 5;10(19):e022515. doi: 10.1161/JAHA.121.022515. Epub 2021 Sep 29. No abstract available. PMID 34585620
- [Background] Lancellotti P, Pibarot P, Chambers J, Edvardsen T, Delgado V, Dulgheru R, Pepi M, Cosyns B, Dweck MR, Garbi M, Magne J, Nieman K, Rosenhek R, Bernard A, Lowenstein J, Vieira ML, Rabischoffsky A, Vyhmeister RH, Zhou X, Zhang Y, Zamorano JL, Habib G. Recommendations for the imaging assessment of prosthetic heart valves: a report from the European Association of Cardiovascular Imaging endorsed by the Chinese Society of Echocardiography, the Inter-American Society of Echocardiography, and the Brazilian Department of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2016 Jun;17(6):589-90. doi: 10.1093/ehjci/jew025. Epub 2016 May 3. PMID 27143783
- [Background] Herrmann HC, Laskey WK. Pressure loss recovery in aortic valve stenosis: Contemporary relevance. Catheter Cardiovasc Interv. 2022 Jan 1;99(1):195-197. doi: 10.1002/ccd.29729. Epub 2021 Apr 22. PMID 33886155
- [Background] Abbas AE, Mando R, Kadri A, Khalili H, Hanzel G, Shannon F, Al-Azizi K, Waggoner T, Kassas S, Pilgrim T, Okuno T, Camacho A, Selberg A, Elmariah S, Bavry A, Ternacle J, Christensen J, Gheewala N, Pibarot P, Mack M. Comparison of Transvalvular Aortic Mean Gradients Obtained by Intraprocedural Echocardiography and Invasive Measurement in Balloon and Self-Expanding Transcatheter Valves. J Am Heart Assoc. 2021 Oct 5;10(19):e021014. doi: 10.1161/JAHA.120.021014. Epub 2021 Sep 29. PMID 34585593
- [Background] Abbas AE, Mando R, Hanzel G, Gallagher M, Safian R, Hanson I, Almany S, Pibarot P, Dalal P, Vivacqua A, Sakwa M, Shannon F. Invasive Versus Echocardiographic Evaluation of Transvalvular Gradients Immediately Post-Transcatheter Aortic Valve Replacement. Circ Cardiovasc Interv. 2019 Jul;12(7):e007973. doi: 10.1161/CIRCINTERVENTIONS.119.007973. Epub 2019 Jul 5. No abstract available. PMID 31272227